CLINICAL TRIAL: NCT05164445
Title: Observational Participants Not Assigned to Intervention(s) Based on a Protocol; Typically in Context of Routine Care
Brief Title: The Role of Interventional Pulmonology, Microbiota and Immune Response in the Patient With Lung Cancer
Acronym: RIPMIRLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Marius Zemaitis, Professor, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RIPMIRLC-001
Record Dates: First submitted 2021-11-18; First posted 2021-12-20 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer
Keywords: cryobiopsy; lung cancer; gut-lung microbiota; immune system
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transbronchial forceps biopsy (Active Comparator): Patients, whose transbronchial forceps biopsy was performed
  Interventions: Diagnostic Test: Transbronchial forceps biopsy
- Transbronchial forceps biopsy+Transbronchial cryobiopsy (Active Comparator): Patients, whose transbronchial forceps biopsy and transbronchial cryobiopsy were performed as well
  Interventions: Diagnostic Test: Transbronchial forceps biopsy+Transbronchial cryobiopsy

INTERVENTIONS:
Diagnostic Test: Transbronchial forceps biopsy — All patients with peripheral lung lesion suspected of lung cancer detected on the chest computed tomography (CT) and mini probe endobronchial ultrasound (RP-EBUS) scans were enrolled. Transbronchial forceps biopsy (TBFB) was performed for all these patients.
  Arms: Transbronchial forceps biopsy
Diagnostic Test: Transbronchial forceps biopsy+Transbronchial cryobiopsy — All patients with peripheral lung lesion suspected of lung cancer detected on the chest computed tomography (CT) and RP-EBUS scans were enrolled. TBFB was performed for all these patients. In addition, all of these patients, with no contraindications, underwent transbronchial cryobiopsy (TBCB)
  Arms: Transbronchial forceps biopsy+Transbronchial cryobiopsy

SUMMARY:
This study is designed to evaluate complications, specificity, diagnostic yield of radial endobronchial ultrasound guided transbronchial cryobiopsy and transbronchial forceps biopsy with fluoroscopy in the diagnosis of peripheral pulmonary lesion; the interplay between non-small-cell lung cancer associated-bacteria along the gut-lung axis and immune response in the cancer microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* patients with peripheral lung lesion suspected of lung cancer detected on the chest computed tomography (CT) and RP-EBUS scans
* Control group - patients without non-small cell lung cancer
* Written (signed) Informed Consent to participate in the study

Exclusion Criteria:

* severe hypoxemia (partial pressure of oxygen (pO2)< 60 mmHg) or hypercapnia (carbon dioxide partial pressure (pCO2)> 50 mmHg),
* bleeding disorders
* The diffusing capacity for carbon monoxide (DLCOc)< 35 %,
* forced expiratory volume in one second (FEV1) < 800 ml or FEV 1 < 30 %,
* peripheral lung tumor was not visualised by RP-EBUS longer than 30 minutes
* large vessels (more than 3 mm) near the tumor on the CT scan,
* technically difficult to introduce cryoprobe and/or endobronchial blocker to current bronchi segment or subsegment,
* excessive bleeding after transbronchial forceps biopsy, which was needed extra intervention to stop bleeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
progression-free survival | one year after enrolment to the study

SECONDARY OUTCOMES:
overall survival | 3 years after enrolment to the study

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania